CLINICAL TRIAL: NCT03062995
Title: A Randomised, Double-blind, Controlled, Parallel-group, Multi-country Study to Investigate the Effect of a Partially Hydrolysed Infant Formula With Added Synbiotics on the Development of Allergic Manifestations in Infants at High Risk of Developing Allergy
Brief Title: A Clinical Study to Investigate the Effect of a Partially Hydrolysed Infant Formula With Added Synbiotics on the Development of Allergic Manifestations in Infants at High Risk of Developing Allergy
Acronym: MAESTRO
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Study design not adequate anymore
Sponsor: Nutricia Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: EBB15BL89859
Record Dates: First submitted 2017-02-01; First posted 2017-02-24 (Actual); Last update posted 2021-12-23 (Actual); Status verified 2021-12

CONDITIONS: Immunity
MeSH Terms: interventions — Infant Formula

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active product: partially hydrolysed formula + synbiotics (Experimental): partially hydrolysed formula + synbiotics
  Interventions: Other: Infant Formula with added synbiotics
- Control product: standard formula (intact protein) (Active Comparator): standard formula (intact protein)
  Interventions: Other: Standard Infant formula

INTERVENTIONS:
Other: Infant Formula with added synbiotics — Intervention group: Infant Formula / Follow-On formula with partially hydrolysed cow's milk protein supplemented with prebiotics and probiotics.
  Arms: Active product: partially hydrolysed formula + synbiotics
Other: Standard Infant formula — Control group: Standard Infant Formula / Follow-On formula with intact cow's milk protein (only standard ingredients, without addition of pre- and probiotics).
  Arms: Control product: standard formula (intact protein)

SUMMARY:
With the rising prevalence of allergic diseases and the subsequent risk of developing other immune-related disorders, primary prevention of allergy has become a major priority. It is generally acknowledged that breastfeeding is one of the main pillars in allergy prevention. Infant formulas based on hydrolysed proteins have been developed to be used by infants at increased risk of developing allergy in case a mother is unable or chooses not to breastfeed her infant. The effect of hydrolysed formula in allergy prevention has been examined in many studies, from which it can be concluded that currently there is not sufficient evidence to support hydrolysed protein over intact protein for allergy risk reduction. Moreover, several clinical trials support the suggestion of supplementation of pre and/or probiotics for the reduction of eczema development, recognized by international authorities. The present study (MAESTRO) investigates the preventive effect of a hypoallergenic concept combining several nutritional approaches related to preventive strategies: partially hydrolysed protein formula supplemented with prebiotics and probiotics. The aim of the present study is to investigate the efficacy, growth and safety of this concept compared to standard (intact protein) infant formula on the development of allergic manifestations up to the age of 12 months in infants at increased risk of developing allergy.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy term infants (gestational age ≥ 37 and ≤ 42 weeks) at high risk of developing allergy based on family history of allergy (*1).
2. Infants aged ≤ 16 weeks (max. 16 weeks + 0 days), preferably as soon as possible after birth.
3. Infants who start formula feeding within 16 weeks of age (infants of mothers who have chosen not to breastfeed or mothers who completely/partially cease breastfeeding before the subject's age of 16 weeks)(*2) OR Infants who are exclusively breastfed and whose mothers have the intention to exclusively breastfeed at least until their infant is 16 weeks of age (*2,3).
4. Written informed consent from one or both parents (according to local laws) and/or legal guardian.

   * 1 Family history of allergy is defined as at least one first-degree relative (parent or full sibling) with: self-reported historically doctor confirmed allergic disease (allergic rhinitis, asthma, food allergy, allergic eczema). In case of a self-reported historically non-doctor confirmed allergic disease doctor confirmation must be done as part of the screening procedure according to local practice (e.g. skin prick test, IgE measurement).
   * 2 Subjects whose mother intents to switch to formula feeding before the subject's age of 16 weeks but in the end still exclusively breastfeed, will be included in the breastfed reference group. The other way around, subjects whose mother intents to exclusively breastfeed for at least 16 weeks, but in the end decides to switch to formula earlier, will be included in the randomised groups. All these subject s should meet all other in-/exclusion criteria.
   * 3 Exclusive breast feeding. WHO definition: only breast milk and no other liquids or solids except for drops or syrups consisting of vitamins, mineral supplements or medicines [2]. In addition to the WHO definition, in this study water is allowed as well as formula feeding during the first 72 hours of life.

Exclusion Criteria:

1. Consumption of any amount of infant formula based on intact protein before randomisation, except for consumption during the first 72 hours of life.
2. Consumption of any amount of infant formula with added probiotics and/or probiotic supplement before randomisation.
3. Existing allergic manifestations (e.g. allergic skin disorders, food allergy) before randomisation according to investigator's clinical assessment.
4. Severe congenital abnormalities which could influence the subjects' growth (e.g. cystic fibrosis, bronchopulmonary dysplasia, tracheomalacia, tracheoesophageal fistula, major congenital heart disease, or any other condition according to investigator's clinical judgement).
5. Severe neonatal illnesses (e.g. respiratory distress syndrome, severe sepsis intraventricular hemorrhage, severe neonatal jaundice, necrotizing enterocolitis, persistent pulmonary hypertension of the newborn, or any other condition which required the use of intravenous and/or intramuscular antibiotics).
6. Known underlying disease predisposing to infection (e.g. HIV, viral hepatitis B, and C, auto-immune diabetes, immune deficiency).
7. Severe renal failure and hepatic failure according to investigator's clinical judgement.
8. Incapability of the parents to comply with study protocol or investigator's uncertainty about the willingness or ability of the subject to comply with the protocol requirements.
9. Participation in other studies involving investigational or marketed products concomitantly or within two weeks prior to screening visit.

Max Age: 16 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2019-06 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Allergic manifestations (IgE-mediated) | 54 weeks
  Doctor diagnosed IgE-mediated allergic manifestations

SECONDARY OUTCOMES:
Allergic manifestations (IgE-mediated and non IgE-mediated) | 54 weeks
  Doctor diagnosed IgE-mediated allergic manifestations and non IgE-mediated allergic manifestations

IPD SHARING:
Plan to Share IPD: No